CLINICAL TRIAL: NCT05598047
Title: Executive Function Training to Reduce Cognitive Intra-Individual Variability in Adults With HIV
Brief Title: Executive Functioning Training Study
Acronym: EFT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, David Vance, PhD, Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB 300008561; 5R21AG077957-02 (NIH)
Record Dates: First submitted 2022-10-13; First posted 2022-10-28 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Aging; Cognitive Function Abnormal; Cognitive Performance; Cognitive Training; Older Adults
MeSH Terms: conditions — Cognition Disorders

STUDY DESIGN:
Intervention Model Description: A pre-post two-group experimental design will be used. One group will receive the experimental executive functioning training and the other group will not receive anything (no-contact control group)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Executive Functioning Training (Experimental): BrainHQ (POSIT Science Inc.) computerized cognitive training modules will be used as in our other studies; but these will focus on executive functioning training. These programs have gaming components that encourage adherence. BrainHQ cognitive training products are tested and endorsed by the scientific community. A meta-analysis of computerized cognitive training in older adults found optimal therapeutic effects occurred when training sessions last at most 60 minutes and are administered 1-3 times per week - dosage parameters already incorporated in our study. This self-administered program uses touch-screen technology with tablets which allows computer novices to engage with the training exercises.
  Interventions: Behavioral: Executive Functioning Training
- No-Contact Control Group (No Intervention): These participants will not receive any intervention.

INTERVENTIONS:
Behavioral: Executive Functioning Training — Those in the Executive Functioning Training Group will engage in exercises requiring one to set shift; that is, to maintain at least two sets of rules and decide which is appropriate to determine the response. In using these training exercises in the TOPS study, the effects size was quite large (d=-0.89). Dosage of 20 hours of training is considered an upper range on how much training is needed to produce an optimal therapeutic effect.
  Arms: Executive Functioning Training

SUMMARY:
Cognitive aging in people with HIV (PWH) is of increasing concern for several reasons: 1) between 52%-59% of PWH experience cognitive impairment known as HIV-Associated Neurocognitive Disorder (HAND) which impacts everyday functioning and quality of life; 2) HAND increases in severity and prevalence with age; and 3) 70% of PWH in the United States will be 50 and older by 2030. Fortunately, cognitive training programs can individually target specific cognitive impairments in PWH and possibly reduce the severity and prevalence of HAND and improve everyday functioning and quality of life. This approach is based around the underlying concept of intra-individual variability as controlled through higher level allocation of cognitive resources, known as executive functioning. This feasibility study will use a two-group pre-post experimental design of adults with HAND including: 1) a 20-hours of Executive Functioning Training group (enroll 60, n=48 with attrition), and 2) a no-contact control (enroll 60, n=48 with attrition). Aim 1 - Feasibility: To determine feasibility and acceptability of the intervention (i.e., attrition, feedback). Exploratory Aim 1 - Cognition: Compare adults who receive Executive Functioning Training to those who receive no training to determine whether they improve in global cognitive ability and overall cognitive IIV. This high impact study is innovative in the following ways: 1) This is the first study aimed to reduce cognitive IIV in PWH. 2) This is the first study to use IIV as a guide to target solely executive functioning training to improve global cognitive ability, which may reduce the severity and prevalence of HAND. 3) Over the last decade, the epicenter of HIV has emerged in the Deep South where this study will occur. Most participants in this study will be older PWH who identify as lower social economic status (SES) and/or African Americans and experience HAND symptoms.

DETAILED DESCRIPTION:
OVERALL -- A pre-post three-group experimental design will be used. Participants will be recruited from the University of Alabama at Birmingham (UAB) 1917 HIV/AIDS Clinic which has a patient population of +3,600 and is the largest HIV medical provider within 100 miles. Eligible participants will be consented at the UAB Center for Research on Applied Gerontology where a ~2 hr baseline assessment will be administered. Participants' neuropsychological data gathered at baseline will be examined to determine a HAND classification. Only participants with HIV-Associated Neurocognitive Disorder (HAND) will be invited to continue with the study. Stratified random assignment will ensure an equal number of participants in each group by gender, minority status, and with/without executive functioning impairment (i.e., 1 standard deviation below normative mean). After training, participants will complete a posttest assessment.

Recruitment/Retention Strategies. As effective in our studies, recruitment/retention strategies will be used. 1) Recruitment materials distributed in the UAB 1917 HIV/AIDS Clinic. 2) Reminder letters and telephone calls will be used before the scheduled visit. 3) Beverages/snacks will be provided (from departmental funds). 5) Secondary contact information will be collected to follow up with lost participants.

Intervention Protocol BrainHQ (POSIT Science Inc.) cognitive training modules will be used as in our other studies; these programs have gaming components that encourage adherence. BrainHQ cognitive training products are tested and endorsed by the scientific community. A meta-analysis of computerized cognitive training in older adults found optimal therapeutic effects occurred when training sessions last at most 60 minutes and are administered 1-3 times per week - dosage parameters already incorporated in our study. This self-administered program uses touch-screen technology with tablets which allows computer novices to engage with the training exercises. The intervention will be administered in the research lab of the UAB Center for Applied Gerontology where many of our other studies have been conducted. Working with BrainHQ, when logging on, participants can only receive the individualized cognitive training exercises they are assigned.

Executive Functioning Training Group. Those in the Executive Functioning Training Group will engage in exercises requiring one to set shift; that is, to maintain at least two sets of rules and decide which is appropriate to determine the response. In using these training exercises in the Training On Purpose Study (TOPS), the effects size was quite large (d=-0.89). Dosage of 20 hours of training is considered an upper range on how much training is needed to produce an optimal therapeutic effect.

No-Contact Control Group. This group will receive no intervention. As this is a pilot/feasibility study, investigators do not have the resources to provide a contact control group. Importantly, in a prior study, investigators established that a no-contact control group and a contact control (sham) group did not significantly differ from each other and both served as an excellent comparison to a cognitive intervention.

Instruments Administration time of the assessment will be ~2 hrs. Investigators will use REDCap and BrainBaseline Assessment of Cognition and Everyday Functioning (BRACE+) tablet for administration of the instruments below to reduce tester burden, tester error, and improve the efficiency of data entry and data management, which will save significant staff time and resources. Other cognitive studies as observed in the HIV Neurobehavioral Research Center (HNRC) group employ testing assessments of similar length. BRACE+ was develop in conjunction with HNRC.

ELIGIBILITY:
Inclusion Criteria:

* Participants (men & women) must be 40+ years
* English speaking,
* Willing to meet in person
* Has time to participate for ~12 weeks

Exclusion Criteria:

* Participants living beyond 60 miles away from the center
* Participants living in unstable housing (e.g., halfway house)
* Participants with significant neuromedical comorbidities (e.g., schizophrenia)
* Participants with other conditions (e.g., legally blind/deaf, currently undergoing radiation or chemotherapy, or a history of significant brain trauma, diagnosed with COVID-19 over the past 3 months) that could impact cognitive functioning or testing.
* Participants who have received cognitive training within the past three years

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2023-06-13 (Actual); Primary Completion 2025-04-08 (Actual); Study Completion 2025-04-08 (Actual)

PRIMARY OUTCOMES:
Baseline Assessment of Cognitive Training | ~12 weeks
  All participants at baseline will be asked questions about computer use, knowledge about cognitive training, their perceptions about whether they need cognitive training, knowledge about HIV and cognition, etc. Both quantitative and qualitative (i.e., open-ended responses) data will be collected; this is similar to our other studies.
Cognitive Training Satisfaction Questionnaire | ~12 weeks
  Used to assess likes/dislikes of the intervention, both quantitative questions and qualitative (i.e., open-ended responses) data are gathered as has been used in our previous cognitive intervention studies to evaluate feasibility and acceptability.
Exit Survey | ~12 weeks
  Investigators will administer a brief quantitative and qualitative (i.e., open-ended responses) survey to assess what he/she liked/disliked about the training and how to improve it.
Adherence Rates (after study data collection) | Through study completion, an average of 2 years
  Investigators will calculate the adherence rate of the protocol, similar to the investigator's other studies. Ranges will be from 0% to 100%.
Attrition Rates (after study data collection) | Through study completion, an average of 2 years
  Investigators will calculate the attrition rate of the protocol, similar to the investigator's other studies. Ranges will be from 0% to 100%.

SECONDARY OUTCOMES:
BRACE+ (BrainBaseline Assessment of Cognition and Everyday Functioning) | ~12 weeks
  Cognitive data will be gathered via BRACE+ (BrainBaseline Assessment of Cognition and Everyday Functioning), supported by NIMH R42099964 and Digital Artefacts/UCSD) is a HIPAA compliant tablet-based cognitive assessment platform. This self-administered tool is not literacy dependent (i.e., automated audio/video instructions) and uses validated cognitive tests sensitive to mild-to-moderate cognitive impairments.

IPD SHARING:
Plan to Share IPD: Yes
We will archive all data electronically without PHI which will be available upon request.
Supporting Information: Study Protocol, SAP
Time Frame: Upon completion of the study
Access Criteria: Based upon IRB approval and Data Use Agreement.

REFERENCES:
- [Background] Vance DE, Fazeli PL, Azuero A, Wadley VG, Raper JL, Ball KK. Can Individualized-Targeted Computerized Cognitive Training Benefit Adults with HIV-Associated Neurocognitive Disorder? The Training on Purpose Study (TOPS). AIDS Behav. 2021 Dec;25(12):3898-3908. doi: 10.1007/s10461-021-03230-y. Epub 2021 Mar 18. PMID 33733311
- [Background] Vance DE, Fazeli PL, Cheatwood J, Nicholson C, Morrison S, Moneyham LD. Targeting HIV-Related Neurocognitive Impairments with Cognitive Training Strategies: Insights from the Cognitive Aging Literature. Curr Top Behav Neurosci. 2021;50:503-515. doi: 10.1007/7854_2018_80. PMID 30710223
- [Background] Waldrop D, Irwin C, Nicholson WC, Lee CA, Webel A, Fazeli PL, Vance DE. The Intersection of Cognitive Ability and HIV: A Review of the State of the Nursing Science. J Assoc Nurses AIDS Care. 2021 May-Jun 01;32(3):306-321. doi: 10.1097/JNC.0000000000000232. PMID 33449578